CLINICAL TRIAL: NCT04995614
Title: The Evaluation of the Health-related Quality of Life, Psychological Distress and Fatigue in Metastatic Castration-resistant Prostate Cancer Patients Treated With Radium-223 Therapy, a Multicenter, Prospective Observational Cohort Study
Brief Title: Health-related Quality of Life, Psychological Distress and Fatigue in Metastatic CRPC Patients Treated With Radium-223
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: AURIMPCA-2; MOURO27 (Other: Radboudumc)
Record Dates: First submitted 2021-07-16; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Castrate Resistant Prostate Cancer; Bone Metastases
Keywords: Radium-223; Health-related quality of life; Psychological distress; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Radium-223; radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Radium-223 — Prospective observational cohort study investigating patient-reported outcomes
  Other Names: Xofigo

SUMMARY:
The aim of the current prospective multicenter study is to evaluate cancer-specific and bone metastases related HR-QoL, psychological distress and fatigue in mCRPC patients before, during and after treatment with radium-223 in daily practice. Furthermore, the investigators aim to determine patient groups with identical health-related quality of life patterns over time, in order to identify variables related to health-related quality of life deterioration during the course of treatment, as patients with health-related quality of life deterioration may need specific attention to preserve health-related quality of life.

DETAILED DESCRIPTION:
Radium-223 is a registered treatment option for patients with symptomatic bone metastatic castration-resistant prostate cancer. Previously, the phase 3 ALSYMPCA trial demonstrated that radium-223 improved overall survival and prolonged the time to the first symptomatic skeletal event and the time to first opioid use, irrespective of prior docetaxel chemotherapy. Subsequent analysis of the ALSYMPCA study showed that a significantly higher percentage of patients receiving radium-223 experienced meaningful HR-QoL improvement, as measured by the EQ-5D questionnaire and the FACT-P questionnaire, when compared to patients treated with placebo. However, studies evaluating health-related quality of life, psychological distress and fatigue in metastatic castration-resistant prostate cancer patients treated with radium-223 in daily practice are lacking.

ELIGIBILITY:
Inclusion criteria:

* Metastatic castration-resistant prostate cancer;
* Undergoing treatment with radium-223 according to standard of care;
* Ability to comply with the study protocol, including completion of questionnaires on health-related quality of life;
* Written informed consent to the treating physician at the hospital site.

Exclusion criteria:

* Prior radium-223 therapy;
* Impaired cognitive functioning and/or illiteracy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastatic castration-resistant prostate cancer patients who are treated with radium-223 in The Netherlands
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Cancer-specific health-related quality of life | 6 months
  Measured with the European Organization for Research and Treatment of Cancer (EORTC) core QoL questionnaire (QLQ-C30). All items are rated on a 4-point Likert-type response scale of 1 ("not at all") to 4 ("very much"), with the exception of the global health status scale items, which are rated from 1-7. Each subscale will be linearly transformed to a 0-100 scale, according to the EORTC scoring manuals. For the functional and global scales, high scores indicate high level of functioning. For the symptom scales, high scores indicate high symptom burden. Clinically relevant changes (CRCs) in EORTC scores are defined as small (5-10 points), moderate (10-20 points), or large (>20 points).
Bone metastases related health-related quality of life | 6 months
  Measured with the European Organization for Research and Treatment of Cancer (EORTC) bone metastases module (BM-22). All items are rated on a 4-point Likert-type response scale of 1 ("not at all") to 4 ("very much"). Each subscale will be linearly transformed to a 0-100 scale, according to the EORTC scoring manuals. For the functional and global scales, high scores indicate high level of functioning. For the symptom scales, high scores indicate high symptom burden. Clinically relevant changes (CRCs) in EORTC scores are defined as small (5-10 points), moderate (10-20 points), or large (>20 points).

SECONDARY OUTCOMES:
Intensity and location of bone pain | at baseline
  Measured with the Brief Pain Inventory Short Form (BPI-SF). The pain severity items are rated on 0-10 scales, with 0 indicating "no pain" and 10 indicating "worst possible pain". Clinically relevant pain is defined as a score of ≥4 on the average pain severity scale.
Psychological distress | 6 months
  Measured with the Hospital Anxiety and Depression Scale (HADS). The HADS contains a 7-item anxiety and a 7-item depression subscale. All items are scored on a 4-point Likert-scale ranging from scores 0 ('never') to 3 ('almost always'). A total score of 11 or higher indicates psychological distress. The clinically relevant chage in HADS subscale scores is defined as 1.5 points change, and 3 points change for the total HADS score.
Fatigue | 6 months
  Measured with the Checklist Individual Strength - Fatigue subscale (CIS-Fatigue). The CIS-Fatigue contains 8 items, and each item is scored on a 7-point Likert scale ranging from "Yes, that is true" to "No, that is not true". A score of 35 or higher on the subscale fatigue severity indicates severe feelings of fatigue.

OTHER OUTCOMES:
Overall survival | 24 months
  Defined as the time between the first radium-223 injection and either death from any cause or the last follow-up
Number of radium-223 injections | 6 months
  Number of radium-223 injections
Trajectory analysis of health-related quality of life patterns over time | 6 months
  Individual responses are classified based upon similar patterns in health-related quality of life, according to the EORTC QLQ-C30 summary score. Summary scores will be classified as <60 (low), 60-80 (intermediate) and >80 (high). Changes in summary scores over time will be classified as deteriorated, stable low (low at all time points), stable intermediate, stable high, improved and fluctuating.

CONTACTS AND LOCATIONS:
Overall Officials: Inge M. van Oort, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (11):
- Netherlands (11):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Ziekenhuisgroep Twente, Almelo
  - Rijnstate ziekenhuis, Arnhem
  - Reinier de Graaf Gasthuis, Delft
  - Catharina ziekenhuis, Eindhoven
  - Universitair medisch centrum Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Canisius-Wilhelmina ziekenhuis, Nijmegen
  - Radboud universitair medisch centrum (Radboudumc), Nijmegen
  - Bravis ziekenhuis, Roosendaal
  - Zuyderland medisch centrum, Sittard

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van der Doelen MJ, Oving IM, Wyndaele DNJ, van Basten JP, Terheggen F, van de Luijtgaarden ACM, Oyen WJG, van Schelven WD, van den Berkmortel F, Mehra N, Janssen MJR, Prins JB, Gerritsen WR, Custers JAE, van Oort IM. Health-related quality of life, psychological distress, and fatigue in metastatic castration-resistant prostate cancer patients treated with radium-223 therapy. Prostate Cancer Prostatic Dis. 2023 Mar;26(1):142-150. doi: 10.1038/s41391-022-00569-8. Epub 2022 Jul 8. PMID 35804188